CLINICAL TRIAL: NCT06866561
Title: The Effect of Aerobic Exercise on Bone Formation and Resorption Markers And The Quality of Life Tests in Postmenopausal Osteopenic Patients
Brief Title: The Effect of Aerobic Exercise on Bone Turnover Markers in Postmenopausal Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bursa Yuksek Ihtisas Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, KÜBRA NUR DENİZ, Principal Investigator, Bursa Yuksek Ihtisas Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HSBY-FTR-KND-01
Record Dates: First submitted 2025-02-20; First posted 2025-03-10 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Postmenopausal Osteopenia
Keywords: postmenopausal osteoporosis; aerobic exercise; bone turnover markers
MeSH Terms: conditions — Osteoporosis, Postmenopausal | interventions — Exercise; Cholecalciferol; Calcium Carbonate

STUDY DESIGN:
Intervention Model Description: Patients who met the inclusion criteria were randomized into 2 groups with the investigator blinded. Participants in the exercise group were included in an aerobic exercise program, while patients in the control group were not included in any exercise program. All patients underwent serum marker assessment and clinical examination both at baseline and after 12 weeks of follow-up.
Who Masked: Investigator
Masking Description: Patients who met the inclusion criteria were randomized into 2 groups with the investigator blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- exercise group (Active Comparator): The exercise group participated in a supervised aerobic exercise program consisting of walking on a treadmill for 30 minutes per day, 3 days per week, at an intensity of 40-60% of maximal heart rate for 4 weeks.
  Interventions: Other: aerobic exercise; Other: cholecalciferol; Other: calcium carbonate
- Control group (Other): The control group did not participate in any exercise program.
  Interventions: Other: cholecalciferol; Other: calcium carbonate

INTERVENTIONS:
Other: aerobic exercise — The exercise group participated in a supervised aerobic exercise program consisting of walking on a treadmill for 30 minutes per day, 3 days per week, at an intensity of 40-60% of maximal heart rate for 4 weeks. Additionally, they were shown an exercise program at the initial assessment that included balance, posture, and endurance exercises using body weight and weights to be performed 3 days a week, with 3 sets of 10 repetitions. The control group did not participate in any exercise program.
  Arms: exercise group
Other: cholecalciferol — Participants were prescribed 2000 IU of vitamin D (cholecalciferol) daily for 12 weeks.
Other: calcium carbonate — Participants were prescribed 1200 mg of calcium carbonate daily for 12 weeks.

SUMMARY:
The aim of the study was to evaluate the effect of light-moderate aerobic exercise on BMD in postmenopausal osteopenic women using bone formation-resorption markers. Participants were randomized into two groups as aerobic exercise and control groups and followed for 12 weeks. At the beginning and at the 12th week, bone formation-resorption markers including procollagen type 1 N-terminal propeptide (P1NP), cross-linked C-telopeptide of type 1 collagen (CTX), osteocalcin, malondialdehyde, non-bone-specific total alkaline phosphatase, 25(OH)D3 and oxidative markers such as parathyroid hormone (PTH) were evaluated in serum and whether there was a difference between the 2 groups.

DETAILED DESCRIPTION:
The aim of the study was to investigate the effects of light and moderate intensity aerobic exercise on bone mineral density (BMD) in postmenopausal osteopenic women using bone formation and resorption markers. In a prospective, randomized, controlled, single-blind clinical trial, women aged 45-65 years with BMD T scores between -1 and -2.5 measured by double X-ray absorptiometry (DXA) were included in the study after evaluation of exclusion criteria and the women were divided into 2 groups: aerobic exercise group and control group (exercise, n=25; control, n=25). The exercise group participated in a supervised aerobic exercise program consisting of walking on a treadmill for 30 minutes per day, 3 days per week, at an intensity of 40-60% of maximal heart rate for 4 weeks. Additionally, they were shown an exercise program at the initial assessment that included balance, posture, and endurance exercises using body weight and weights to be performed 3 days a week, with 3 sets of 10 repetitions. The control group did not participate in any exercise program.All patients were prescribed 2000 IU of vitamin D (cholecalciferol) and 1200 mg of calcium carbonate daily for 12 weeks. Serum levels of biomarkers of bone formation and resorption including procollagen type 1 N-terminal propeptide (P1NP), cross-linked C-telopeptide of type 1 collagen (CTX), osteocalcin, malondialdehyde, non-bone-specific total alkaline phosphatase, 25(OH)D3 and oxidative markers such as parathyroid hormone (PTH) were examined in all patients at baseline and 12-week follow-up. Nottingham Health Profile questionnaire (NHP), Visual analog scale (VAS), 6-minute walk test (6MWT), International Physical Activity Questionnaire (short form) (IPAQ), Berg Balance Scale (BBS), 30-second sit-to-stand test questionnaires (30s-CST) tests were performed at baseline and 12 weeks to evaluate the participants' quality of daily life, pain, walking speed, physical activity level and balance.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women from Türkiye aged 45-65 years,
* Bone mineral density (BMD) T-scores between -1 and -2.5 ( measured by dual-energy X-ray absorptiometry)

Exclusion Criteria:

* Vertebral compression fracture,
* A history of traumatic or nontraumatic fractures in the past year,
* Thyroid hormone disorders,
* Parathyroid hormone disorders,
* Liver function disorders,
* Kidney function disorders,
* Chronic heart failure,
* A history of malignancy,
* A history of rheumatological diseases,
* Corticosteroid use,
* Immunosuppressive drug use,
* Anticonvulsant and heparin use,
* Antiresorptive or anabolic agent treatments use
* Hormone replacement therapy use
* Those who could not complete sessions due to mechanical pain exacerbated during aerobic exercise on a treadmill (such as knee and hip osteoarthritis, back pain, etc)

Ages: 45 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2022-11-15 (Actual); Primary Completion 2023-11-15 (Actual); Study Completion 2023-11-15 (Actual)

PRIMARY OUTCOMES:
The serum levef of Procollagen type 1 N-terminal propeptide (P1NP) (ng/ml) | From enrollment to the end of treatment at 12 weeks
  Bone turnover markers allow for the independent assessment of bone resorption and formation by measuring their concentrations in blood and urine. These markers provide early response evaluation posttreatment of osteoporosis compared to measuring BMD. The International Osteoporosis Foundation (IOF) and the International Federation of Clinical Chemistry and Laboratory Medicine (IFCC) recommend evaluating P1NP for bone formation activity and evaluating CTX-1 concentrations for bone resorption activity. In the study,the investigators chose walking exercise as an aerobic exercise that can be easily applied to people of all age groups and those with comorbidities. For these reasons, as the primary outcome of the study, the investigators aimed to measure the effects of aerobic exercise as a treatment method that can be recommended to the majority of patients, as bone turnover markers P1NP, CTX, OCN and total ALP respond quickly to treatment.
The serum levef of Cross-linked C-telopeptide of type I collagen (CTX) (ng/ml) | From enrollment to the end of treatment at 12 weeks
  During bone resorption, components of bone tissue are catabolized by osteoclasts. The released components are released into the bone microenvironment and secreted into the bloodstream. Some of them are also excreted in the urine. The level of C-telopeptide type 1 collagen(CTX)(ng/ml) can be measured in serum from these products. . The International Osteoporosis Foundation (IOF) and the International Federation of Clinical Chemistry and Laboratory Medicine (IFCC) recommend evaluating CTX-1 concentrations for bone resorption activity.
The serum levef of Osteocalcin(OCN) (ng/ml) | From enrollment to the end of treatment at 12 weeks
  During bone formation, osteoblasts fill the cavities with collagen-rich tissue and the molecules formed during their production are secreted into the blood. These products are; Type 1 procollagen N-terminal propeptide (P1NP), bone alkaline phosphatase, Osteocalcin, Type-1 procollagen C-terminal propeptide. These molecules also show bone formation activity.
The serum levef of nonbone-specific total alkaline phosphatase (ALP) (U/L) | From enrollment to the end of treatment at 12 weeks
  During bone formation, osteoblasts fill the cavities with collagen-rich tissue and the molecules formed during their production are secreted into the blood. These products are; Type 1 procollagen N-terminal propeptide (P1NP), bone alkaline phosphatase, Osteocalcin, Type-1 procollagen C-terminal propeptide. These molecules also show bone formation activity.

SECONDARY OUTCOMES:
Serum level of Malondİaldehyde(MDA) (ng/ml) as a Oxidative stress marker | From enrollment to the end of treatment at 12 weeks
  Oxidative stress is considered an important pathogenic factor of osteoporosis at the cellular and molecular level. It induces osteocyte apoptosis and altered levels of specific factors such as receptor activator κB ligand (RANKL), sclerostin and fibroblast growth factor 23, leading to impaired bone remodeling and increased bone resorption. Increased osteoclastic activity occurring in osteoporosis results in increased production of ROS in the form of superoxide. Lipid peroxidation is one of the most deleterious effects of ROS, and the end product of lipid peroxidation, malondialdehyde (MDA), also serves as a measure of osteoclastic activity. For this reason, increased levels of MDA as a marker of oxidative stress can be detected in individuals with osteoporosis. In the study, the investigators aimed to observe the changes in the serum level of malondialdehyde, one of the oxidative stress markers, with aerobic exercise.
Nottingham Health Profile questionnaire (NHP) | From enrollment to the end of treatment at 12 weeks
  Nottingham Health Profile questionnaire (NHP) was used to measure patients' quality of life. NHP consists of section 1 consisting of 38 detailed questions about health and section 2 consisting of 7 questions about the areas of daily life most affected by health. Section 1 questions 6 areas related to health in detail: pain, emotional reactions, sleep, social isolation, physical activity, energy. Each subsection is evaluated between 0-100 points. Section 2 consists of seven statements about the areas of daily life most affected by health: work, daily chores at home, social life, personal relationships, sexual life, hobbies-interests, and holidays. Here, patients are evaluated between 0-7 points, with 1 point for each statement. Patients were evaluated between 0-600 points for section 1, 0-7 points for section 2, and 0-607 points as the NHP Total score.
Visual analog scale (VAS) | From enrollment to the end of treatment at 12 weeks
  Visual analog scale (VAS) was used to evaluate and monitor the level of pain felt by the patients. The investigators aimed to evaluate the pain level of patients after exercise with VAS.Patients were asked to mark on a 100 mm long line divided into 10 units and numbered from 0 to 10; 0 (zero) "I have no pain", 10 "the most severe pain I have ever felt". The number marked was recorded as the VAS pain score.
6-minute walk test (6MWT) | From enrollment to the end of treatment at 12 weeks
  6-minute walk test (6MWT) was used to assess the functional capacity of patients and is a valid and reliable test as an indicator of physical endurance in elderly individuals. The investigators aimed to evaluate the functional capacity of patients after exercise with 6MWT.
International Physical Activity Questionnaire (short form)(IPAQs) | From enrollment to the end of treatment at 12 weeks
  The International Physical Activity Questionnaire (short form) (IPAQs) is used to assess daily physical activity levels. IPAQs consist of 7 questions that assess the time patients spent physically in the last 7 days. These questions assess physical activity in 2 categories: vigorous, moderate and low-level physical activity or weekly MET/minute. MET/minute indicates the amount of energy expended while performing physical activity. While IPAQs are calculated as weekly METs, 3.3 METs are calculated for a minute of low-level physical activity; 4 METs for moderate-level physical activities; 8 METs for a minute of vigorous physical activities. Expending 1500-3000 METs of energy in 1 week is considered vigorous physical activity; 600-1500 METs is considered moderate physical activity, and individuals with less than 600 METs are considered in the light physical activity group. The investigators aimed to assess participants' post-exercise physical activity levels with IPAQs.
Berg Balance Scale (BBS) | From enrollment to the end of treatment at 12 weeks
  Berg Balance Scale (BBS) is a 14-question test used to evaluate the balance and fall risk of elderly individuals. Each item is scored between 0-4 according to the patient's level and speed of performing the desired movement. Patients were evaluated between 0-56 points in total. 0-20 points indicate balance disorder, 21-40 points indicate acceptable balance, and 41-56 points indicate good balance. The investigators aimed to evaluate the balance level of patients after exercise with BBS.
30-second sit-to-stand test questionnaires(30s-CST) | From enrollment to the end of treatment at 12 weeks
  30-second sit-to-stand test questionnaires(30s-CST) evaluates the patient's lower extremity strength and dynamic balance during activity. The investigators aimed to evaluate the lower extremity strength and dynamic balance of the patients after exercise.
The serum levef of Parathyroid hormone (PTH)(pg/ml) | From enrollment to the end of treatment at 12 weeks
  Parathyroid hormone (PTH) plays an important role in regulating calcium and phosphorus metabolism in the body by acting directly on human bones and kidneys and indirectly on the human intestine. In doing so, it affects both bone formation and bone resorption.

CONTACTS AND LOCATIONS:
Overall Officials: Kübra Nur Deniz, M.D., Principal Investigator — Bursa Yuksek Ihtisas Training and Research Hospital
Locations (1):
- Bursa Yüksek İhtisas Education and Research Hospital, Bursa, Yıldırım, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The datasets used and/or analyzed during the current study are provided within the manuscript and supplementary information file.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: The IPD and additional supporting information will be available for sharing 3 months after the study is published.

REFERENCES:
- [Result] Zhou Q, Zhu L, Zhang D, Li N, Li Q, Dai P, Mao Y, Li X, Ma J, Huang S. Oxidative Stress-Related Biomarkers in Postmenopausal Osteoporosis: A Systematic Review and Meta-Analyses. Dis Markers. 2016;2016:7067984. doi: 10.1155/2016/7067984. Epub 2016 Aug 10. PMID 27594735
- [Result] Voulgaridou G, Papadopoulou SK, Detopoulou P, Tsoumana D, Giaginis C, Kondyli FS, Lymperaki E, Pritsa A. Vitamin D and Calcium in Osteoporosis, and the Role of Bone Turnover Markers: A Narrative Review of Recent Data from RCTs. Diseases. 2023 Feb 8;11(1):29. doi: 10.3390/diseases11010029. PMID 36810543
- [Result] Eastell R, Garnero P, Audebert C, Cahall DL. Reference intervals of bone turnover markers in healthy premenopausal women: results from a cross-sectional European study. Bone. 2012 May;50(5):1141-7. doi: 10.1016/j.bone.2012.02.003. Epub 2012 Feb 12. PMID 22348982
- [Result] Siwapituk W, Kitisomprayoonkul W. Bone turnover increases during supervised treadmill walking in Thai postmenopausal women. Osteoporos Sarcopenia. 2016 Mar;2(1):41-44. doi: 10.1016/j.afos.2016.02.005. Epub 2016 Mar 21. PMID 30775467
- [Result] FilipoviC TN, LazoviC MP, BackoviC AN, FilipoviC AN, IgnjatoviC AM, DimitrijeviC SS, GopCeviC KR. A 12-week exercise program improves functional status in postmenopausal osteoporotic women: randomized controlled study. Eur J Phys Rehabil Med. 2021 Feb;57(1):120-130. doi: 10.23736/S1973-9087.20.06149-3. Epub 2020 Sep 9. PMID 32902207
- [Result] Hettchen M, von Stengel S, Kohl M, Murphy MH, Shojaa M, Ghasemikaram M, Bragonzoni L, Benvenuti F, Ripamonti C, Benedetti MG, Julin M, Risto T, Kemmler W. Changes in Menopausal Risk Factors in Early Postmenopausal Osteopenic Women After 13 Months of High-Intensity Exercise: The Randomized Controlled ACTLIFE-RCT. Clin Interv Aging. 2021 Jan 11;16:83-96. doi: 10.2147/CIA.S283177. eCollection 2021. PMID 33469276
- [Result] Zhang L, Zheng YL, Wang R, Wang XQ, Zhang H. Exercise for osteoporosis: A literature review of pathology and mechanism. Front Immunol. 2022 Sep 9;13:1005665. doi: 10.3389/fimmu.2022.1005665. eCollection 2022. PMID 36164342
- [Result] Cariati I, Bonanni R, Onorato F, Mastrogregori A, Rossi D, Iundusi R, Gasbarra E, Tancredi V, Tarantino U. Role of Physical Activity in Bone-Muscle Crosstalk: Biological Aspects and Clinical Implications. J Funct Morphol Kinesiol. 2021 Jun 21;6(2):55. doi: 10.3390/jfmk6020055. PMID 34205747
- [Result] Shoback D, Rosen CJ, Black DM, Cheung AM, Murad MH, Eastell R. Pharmacological Management of Osteoporosis in Postmenopausal Women: An Endocrine Society Guideline Update. J Clin Endocrinol Metab. 2020 Mar 1;105(3):dgaa048. doi: 10.1210/clinem/dgaa048. PMID 32068863
- [Result] Eriksen EF. Treatment of osteopenia. Rev Endocr Metab Disord. 2012 Sep;13(3):209-23. doi: 10.1007/s11154-011-9187-z. PMID 21710179
- [Result] Kaplan AA. A simple and accurate method for prescribing plasma exchange. ASAIO Trans. 1990 Jul-Sep;36(3):M597-9. PMID 2252761
- [Result] Price DD, McGrath PA, Rafii A, Buckingham B. The validation of visual analogue scales as ratio scale measures for chronic and experimental pain. Pain. 1983 Sep;17(1):45-56. doi: 10.1016/0304-3959(83)90126-4. PMID 6226917
- [Result] Hunt SM, McEwen J, McKenna SP. Measuring health status: a new tool for clinicians and epidemiologists. J R Coll Gen Pract. 1985 Apr;35(273):185-8. PMID 3989783
- [Result] Kucukdeveci AA, McKenna SP, Kutlay S, Gursel Y, Whalley D, Arasil T. The development and psychometric assessment of the Turkish version of the Nottingham Health Profile. Int J Rehabil Res. 2000 Mar;23(1):31-8. doi: 10.1097/00004356-200023010-00004. PMID 10826123
- [Result] Yang S, Feskanich D, Willett WC, Eliassen AH, Wu T. Association between global biomarkers of oxidative stress and hip fracture in postmenopausal women: a prospective study. J Bone Miner Res. 2014 Dec;29(12):2577-83. doi: 10.1002/jbmr.2302. PMID 24957524
- [Result] Zhao F, Guo L, Wang X, Zhang Y. Correlation of oxidative stress-related biomarkers with postmenopausal osteoporosis: a systematic review and meta-analysis. Arch Osteoporos. 2021 Jan 5;16(1):4. doi: 10.1007/s11657-020-00854-w. PMID 33400044
- [Result] Marcucci G, Domazetovic V, Nediani C, Ruzzolini J, Favre C, Brandi ML. Oxidative Stress and Natural Antioxidants in Osteoporosis: Novel Preventive and Therapeutic Approaches. Antioxidants (Basel). 2023 Feb 3;12(2):373. doi: 10.3390/antiox12020373. PMID 36829932
- [Result] Vasikaran S, Cooper C, Eastell R, Griesmacher A, Morris HA, Trenti T, Kanis JA. International Osteoporosis Foundation and International Federation of Clinical Chemistry and Laboratory Medicine position on bone marker standards in osteoporosis. Clin Chem Lab Med. 2011 Aug;49(8):1271-1274. doi: 10.1515/CCLM.2011.602. Epub 2011 May 24. PMID 21605012
- [Result] Mohr M, Helge EW, Petersen LF, Lindenskov A, Weihe P, Mortensen J, Jorgensen NR, Krustrup P. Effects of soccer vs swim training on bone formation in sedentary middle-aged women. Eur J Appl Physiol. 2015 Dec;115(12):2671-9. doi: 10.1007/s00421-015-3231-8. Epub 2015 Aug 9. PMID 26255288
- [Result] Jain S, Camacho P. Use of bone turnover markers in the management of osteoporosis. Curr Opin Endocrinol Diabetes Obes. 2018 Dec;25(6):366-372. doi: 10.1097/MED.0000000000000446. PMID 30299435
- [Result] Lorentzon M, Branco J, Brandi ML, Bruyere O, Chapurlat R, Cooper C, Cortet B, Diez-Perez A, Ferrari S, Gasparik A, Herrmann M, Jorgensen NR, Kanis J, Kaufman JM, Laslop A, Locquet M, Matijevic R, McCloskey E, Minisola S, Pikner R, Reginster JY, Rizzoli R, Szulc P, Vlaskovska M, Cavalier E. Algorithm for the Use of Biochemical Markers of Bone Turnover in the Diagnosis, Assessment and Follow-Up of Treatment for Osteoporosis. Adv Ther. 2019 Oct;36(10):2811-2824. doi: 10.1007/s12325-019-01063-9. Epub 2019 Aug 22. PMID 31440982
- [Result] Greenblatt MB, Tsai JN, Wein MN. Bone Turnover Markers in the Diagnosis and Monitoring of Metabolic Bone Disease. Clin Chem. 2017 Feb;63(2):464-474. doi: 10.1373/clinchem.2016.259085. Epub 2016 Dec 9. PMID 27940448
- [Result] Eastell R, Szulc P. Use of bone turnover markers in postmenopausal osteoporosis. Lancet Diabetes Endocrinol. 2017 Nov;5(11):908-923. doi: 10.1016/S2213-8587(17)30184-5. Epub 2017 Jul 7. PMID 28689768
- [Result] Howe TE, Shea B, Dawson LJ, Downie F, Murray A, Ross C, Harbour RT, Caldwell LM, Creed G. Exercise for preventing and treating osteoporosis in postmenopausal women. Cochrane Database Syst Rev. 2011 Jul 6;2011(7):CD000333. doi: 10.1002/14651858.CD000333.pub2. PMID 21735380
- [Result] Todd JA, Robinson RJ. Osteoporosis and exercise. Postgrad Med J. 2003 Jun;79(932):320-3. doi: 10.1136/pmj.79.932.320. PMID 12840119
- [Result] Benedetti MG, Furlini G, Zati A, Letizia Mauro G. The Effectiveness of Physical Exercise on Bone Density in Osteoporotic Patients. Biomed Res Int. 2018 Dec 23;2018:4840531. doi: 10.1155/2018/4840531. eCollection 2018. PMID 30671455
- [Result] NIH Consensus Development Panel on Osteoporosis Prevention, Diagnosis, and Therapy. Osteoporosis prevention, diagnosis, and therapy. JAMA. 2001 Feb 14;285(6):785-95. doi: 10.1001/jama.285.6.785. PMID 11176917
- [Result] Tu KN, Lie JD, Wan CKV, Cameron M, Austel AG, Nguyen JK, Van K, Hyun D. Osteoporosis: A Review of Treatment Options. P T. 2018 Feb;43(2):92-104. PMID 29386866
- [Result] Consensus development conference: diagnosis, prophylaxis, and treatment of osteoporosis. Am J Med. 1993 Jun;94(6):646-50. doi: 10.1016/0002-9343(93)90218-e. No abstract available. PMID 8506892
- [Derived] Deniz KN, Aksoy MK. "The effect of aerobic exercise on bone formation and resorption markers and the quality of life tests in postmenopausal osteopenic patients". BMC Musculoskelet Disord. 2025 Apr 21;26(1):385. doi: 10.1186/s12891-025-08578-z. PMID 40259282

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-12-23): https://cdn.clinicaltrials.gov/large-docs/61/NCT06866561/Prot_SAP_000.pdf